CLINICAL TRIAL: NCT03750851
Title: CPP-ACPF and Low Level Laser Therapy Effect on Symptomatology and Quality of Life of People With Dentin Hypersensitivity: A Clinical, Randomized, Double-blind Study
Brief Title: CPP-ACPF and Laser's Effect on Dentin Hypersensitivity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal do Para (Other)
Responsible Party: Principal Investigator, Cecy Martins Silva, PhD Clinical Professor, Universidade Federal do Para
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UFPara-005
Record Dates: First submitted 2018-11-19; First posted 2018-11-23 (Actual); Last update posted 2019-04-17 (Actual); Status verified 2019-04

CONDITIONS: Dentin Sensitivity
Keywords: desensitizing treatment; dental hypersensitivity; CPPACPF; Low level laser therapy
MeSH Terms: conditions — Dentin Sensitivity | interventions — Lasers

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- GPlacebo (Placebo Comparator): In this group, a water soluble gel without addition any desensitizing agent (K-Y®, Johnson & Johnson, Brazil) was applied to hypersensitive dentin. The GPlacebo volunteers were submitted to the application of placebo dentifrice on the vestibular surfaces of hypersensitive teeth with the aid of a microbrush applicator (Microbrush, 3M ESPE, Brazil) and left undisturbed on the surface during 05 minutes. Then, a rubber cup (Unid Microdont, Brazil) mounted on a low speed handpiece (500, Kavo, Germany) was used to scrub the placebo gel for 20 seconds on each tooth.
  Interventions: Other: Placebo
- GCPPACPF (Experimental): In this group, a toothpaste MI Paste Plus™ (Recaldent™, GC América, USA) was applied to hypersensitive dentin. The GCPPACPF volunteers were submitted to the application of the paste dentifrice on the vestibular surfaces of hypersensitive teeth with the aid of a microbrush applicator (Microbrush, 3M ESPE, Brazil) and left undisturbed on the surface during 05 minutes. Then, a rubber cup (Unid Microdont, Brazil) mounted on a low speed handpiece (500, Kavo, Germany) were used to scrub the desensitizing gel for 20 seconds on each tooth.
  Interventions: Other: CPPACPF
- GLaser (Experimental): In this group, the diode laser with an active medium of Asauxa bauxite (Photon Lase III, DMC Equipamentos Ltda, Brazil) was applied in hypersensitive dentin. GLaser received the laser application using the infrared light spectrum with wavelength of 808 nm with its active AsGaAl medium in two points of the vestibular face of the hypersensitive teeth. It was applied at each point 60 J / cm², for 16 seconds. The laser was applied in 3 sessions with a time interval of 24 hours between them.
  Interventions: Other: Laser
- GLaserCPPACPF (Experimental): In this group the laser + CPP-ACPF was applied. The laser was used with light intensity medium Asauxa (Photon Lase III, DMC Equipamentos Ltda, Brazil) and a toothpaste containing CPP-ACPF MI Paste Plus™ (Recaldent™, GC América, USA) was applied in hypersensitive dentin. GLaserCPPacpf first named a toothpaste application and them the laser application, according to the manufacturer's recommendations.
  Interventions: Other: LaserCPPACPF

INTERVENTIONS:
Other: Placebo — In this group, a water soluble gel without addition any desensitizing agent (K-Y®, Johnson & Johnson, Brazil) was applied to hypersensitive dentin. The GPlacebo volunteers were submitted to the application of placebo dentifrice on the vestibular surfaces of hypersensitive teeth with the aid of a microbrush applicator (Microbrush, 3M ESPE, Brazil) and left undisturbed on the surface during 05 minutes. Then, a rubber cup (Unid Microdont, Brazil) mounted on a low speed handpiece (500, Kavo, Germany) was used to scrub the placebo gel for 20 seconds on each tooth.
  Arms: GPlacebo
Other: CPPACPF — In this group, a toothpaste MI Paste Plus™ (Recaldent™, GC América, USA) was applied to hypersensitive dentin. The GCPPACPF volunteers were submitted to the application of the paste dentifrice on the vestibular surfaces of hypersensitive teeth with the aid of a microbrush applicator (Microbrush, 3M ESPE, Brazil) and left undisturbed on the surface during 05 minutes. Then, a rubber cup (Unid Microdont, Brazil) mounted on a low speed handpiece (500, Kavo, Germany) were used to scrub the desensitizing gel for 20 seconds on each tooth.
  Arms: GCPPACPF
Other: Laser — In this group, the diode laser with an active medium of Asauxa bauxite (Photon Lase III, DMC Equipamentos Ltda, Brazil) was applied in hypersensitive dentin. GLaser received the laser application using the infrared light spectrum with wavelength of 808 nm with its active AsGaAl medium in two points of the vestibular face of the hypersensitive teeth. It was applied at each point 60 J / cm², for 16 seconds. The laser was applied in 3 sessions with a time interval of 24 hours between them.
  Arms: GLaser
Other: LaserCPPACPF — In this group the laser + CPP-ACPF was applied. The laser was used with light intensity medium Asauxa (Photon Lase III, DMC Equipamentos Ltda, Brazil) and a toothpaste containing CPP-ACPF MI Paste Plus™ (Recaldent™, GC América, USA) was applied in hypersensitive dentin. GLaserCPPacpf first named a toothpaste application and them the laser application, according to the manufacturer's recommendations.
  Arms: GLaserCPPACPF

SUMMARY:
The aim of this study was to evaluate the effect of casein phosphopeptide amorphous calcium phosphate fluoride paste (CPP-ACPF) associated with low level laser therapy (LLLT) in the symptomatology and on the quality of life of the individuals with dentin hypersensitivity in a randomized placebo-controlled clinical trial. Volunteers 18 to 50 years old with hypersensitive teeth were randomized into 4 groups: GPlacebo - positioning of the laser tip without light emission + placebo dentifrice; GCPPACPF - positioning of the laser tip without light emission + CPP-ACPF application; GLaser - laser tip positioning with light emission + placebo dentifrice; GLaserCPPACPF - positioning and light emission of the laser beam + CPP-ACPF.

DETAILED DESCRIPTION:
GLaser received the laser application using the infrared light spectrum with wavelength of 808 nm with its active AsGaAl medium in two points of the vestibular face of the hypersensitive teeth. At each point it was applied 60 J / cm², for 16 seconds. Three laser's sessions were applied with a time interval of 24 hours between them. GLaserCPPACPF first received the CPPACPF application and then the laser application according to the manufacturer's recommendations. Before initiating laser therapy, the equipment was calibrated with a tester (MMOptics Ltda®, Brazil).

The GCPPACPF volunteers were submitted to the application of the CPPACPF'S containing tooth paste MI Paste Plus™ (Recaldent™, GC América, USA) on the vestibular surfaces of hypersensitive teeth with the aid of a microbrush applicator (Microbrush, 3M ESPE, Brazil) for 05 minutes. Then, a rubber cup (Unid Microdont, Brazil) mounted on a low speed handpiece (500, Kavo, Germany) was used to scrub the desensitizing gel during 20 seconds on each tooth, according to the manufacturer's specifications. GPlacebo followed the same protocol used in GCPPACPF. In addition to the desensitizing treatments, all GCPPACPF and GPlacebo volunteers received the positioning of the laser tip to mimic the light emission produced in GLaser and GLaserCPPACPF. The noise emitted by the laser device was mimic through the sound reproduction of a smartphone application (HD Voice Recorder - iPhone 6s, Apple®, USA).

ELIGIBILITY:
Inclusion Criteria:

* The presence of at least two hypersensitive teeth;

Exclusion Criteria:

* Milk's proteins allergy;
* Systemic diseases;
* Teeth with carious lesions or pulpitis;
* Teeth with defective restorations;
* Teeth with with cleft enamel;
* Patients with active periodontal disease;
* Patients with analgesic medication;
* Patients with pregnant or lactating women
* Patients who have received professional desensitizing treatment in the last three months.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2018-06-11 (Actual); Primary Completion 2018-12-07 (Actual); Study Completion 2018-12-14 (Actual)

PRIMARY OUTCOMES:
Efficacy of treatment in dental sensitivity intensity change as assessed by VAS | 1 month
  Self reported dentin sensitivity intensity before and after desensitizing treatment. Giving an score for each tooth by marking in the Visual Analogue Scale (VAS) from 0-10 (0-no pain and 10-pain as bad as it can be). With lower values representing a better outcome.
Quality of life change | 1 month
  Self reported dentin sensitivity intensity impact in the quality's of life before and after desensitizing treatment. By answering an specific questionnaire: Dentine Hypersensitivity Experience Questionnaire, measured in a likert scale from 7 to 1 (Where 7 is strongly agree and 1 is strongly disagree). With lower values representing a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Cecy M Silva, PhD, Principal Investigator — clinical professor
Locations (1):
- Para's Federal University, Belém, Pará, Brazil

IPD SHARING:
Plan to Share IPD: Undecided